CLINICAL TRIAL: NCT06762782
Title: Clinical Study on the Effectiveness and Safety of Lenvatinib As Adjuvant Treatment for Patients with High-risk Recurrence of Hepatocellular Carcinoma After Surgery
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: The First People's Hospital of Changzhou (Other); Affiliated Hospital of Nantong University (Other); Suzhou Municipal Hospital (Other); Zhongda Hospital (Other); Northern Jiangsu People's Hospital (Other); The First People's Hospital of Lianyungang (Other); The Affiliated Hospital of Xuzhou Medical University (Other); Xuzhou Central Hospital (Other); Huai'an First People's Hospital (Other); Jiangsu Taizhou People's Hospital (Other)
Responsible Party: Principal Investigator, Haomin Zhou, Professor, The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-SR-708
Record Dates: First submitted 2024-12-22; First posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2024-12

CONDITIONS: Hepatocellular Carcinoma (HCC); Adjuvant Therapy in Patients with Hepatocellular Carcinoma (HCC) At High Risk of Recurrence After Curative Resection or Ablation
Keywords: lenvatinib；adjuvant therapy；hepatocellular carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Intervention Model Description: Eligible subjects were randomly assigned to the experimental group or the control group at a ratio of 2:1, with surgical method (radical surgery vs ablation) as the stratification factor.
  Treatment group:
  According to the instructions, lenvatinib 8mg (weight ≤ 60Kg) or 12mg (weight ≥ 60Kg) was given orally once a day, and active monitoring was performed.
  Control group:
  After surgery, the best supportive care was given, and active monitoring was performed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment group (Experimental): According to the instructions, lenvatinib 8mg (weight ≤ 60Kg) or 12mg (weight ≥ 60Kg) was given orally once a day, and active monitoring was performed.
  Interventions: Drug: Postoperative adjuvant lenvatinib
- Control group (Other): After surgery, the best supportive care was given, and active monitoring was performed.
  Interventions: Other: Supportive care measures

INTERVENTIONS:
Drug: Postoperative adjuvant lenvatinib — Follow the instructions and take lenvatinib 8 mg (body weight ≤ 60Kg) or 12 mg (body weight ≥ 60Kg) orally once a day.
  Arms: Treatment group
Other: Supportive care measures — Adjuvant treatments such as antiviral, TACE, HAIC, radiotherapy, and systemic antitumor therapy can be used
  Arms: Control group

SUMMARY:
This study is a prospective, randomized, controlled, open, phase II, multicenter clinical study, which aims to evaluate the efficacy and safety of lenvatinib for adjuvant treatment of high-risk recurrent liver cancer after radical surgery.

This study is divided into 3 stages: screening period (screening period 28 days), treatment period (up to 12 months, or until any of the following occurs, whichever occurs first: ① The subject has an intolerable toxic reaction and is still not relieved after dose adjustment; ② The subject's first imaging confirmed disease recurrence or withdrew from the study for other reasons), and follow-up period (12 months after the end of treatment).

Dosage regimen:

Eligible subjects were randomly assigned to the experimental group or the control group in a 2:1 ratio, with surgical method (radical surgery vs ablation) as the stratification factor. The experimental group received lenvatinib treatment, and the control group received best supportive care

ELIGIBILITY:
Inclusion Criteria:

* Certainly, here is the translation of the provided text into English:

  1. Age between 18 to 80 years old, gender not limited;
  2. Received radical treatment surgery for liver cancer within 4 to 8 weeks prior to enrollment, and meet the following criteria: (1) Intraoperative judgment criteria: ① No gross tumor thrombus in the hepatic vein, portal vein, bile duct, and inferior vena cava; ② No invasion of adjacent organs, no hepatic hilum lymph nodes or distant metastasis; ③ The liver resection margin is ≥1cm from the tumor border; if the margin is less than 1cm, the histological examination of the resected liver surface shows no residual tumor cells, i.e., negative resection margin. (2) Postoperative judgment criteria: ① Ultrasound, computed tomography(CT), magnetic resonance imaging(MRI) examinations (at least two of these) are performed within 1 to 2 months after surgery, with no residual or recurrent tumor lesions in radical resection cases, and no active tumor lesions in radical ablation cases; ② If serum alpha-fetoprotein(AFP), des-gamma-carboxy prothrombin(DCP), and a combination of 7 Micro ribonucleic acid(microRNAs) and other tumor markers were elevated before surgery, then quantitative measurement of tumor markers is required 8 weeks after surgery, and their levels drop to the normal range; if serum alpha-fetoprotein(AFP) does not return to normal within 8 weeks after surgery , will not be included.
  3. Postoperative pathological examination confirms hepatocellular carcinoma(HCC), and all tumor nodules are completely removed with negative resection margins.
  4. Imaging examinations ≥4 weeks after surgery confirm no recurrence or metastasis.
  5. Expected survival >3 months;
  6. hepatitis B virus(HBV) deoxyribonucleic acid(DNA) <10^4 copies/ml (2000 IU/ml), if hepatitis B virus(HBV) deoxyribonucleic acid(DNA) ≥10^4 copies/ml, antiviral treatment should be initiated first until hepatitis B virus(HBV) deoxyribonucleic acid(DNA) is reduced to below 10^4 copies/ml before entering the study, and continue to take antiviral medication and monitor liver function and hepatitis B virus(HBV) load.
  7. At least one of the following high recurrence risk factors exists:

  <!-- -->

  1. Tumor diameter >5cm
  2. Multiple lesions (>3)
  3. Pathology indicates MVI positivity
  4. Edmondson III-IV grade
  5. Persistently abnormal alpha-fetoprotein 8. No history of other tumors, and no antitumor treatment before surgery; 9. Eastern Cooperative Oncology Group(ECOG) score: 0-1. 10. Major organ functions are normal, i.e., meeting the following criteria:

Hematology examination (within 14 days before screening, without blood transfusion or use of granulocyte colony stimulating factor(G-CSF)):

1. Hemoglobin ≥90 g/L;
2. Absolute neutrophil count (ANC) ≥1.5×10^9/L;
3. Platelet count ≥75×10^9/L;

   Biochemical examination (within 14 days before screening, without the use of albumin):
4. Albumin ≥28 g/L;
5. Total bilirubin ≤1.5×upper limit of normal (ULN);
6. Aspartate aminotransferase (AST), Alanine aminotransferase (ALT) ≤3×ULN;
7. Creatinine ≤1.5×ULN;

   Coagulation function:
8. International normalized ratio (INR) or prothrombin time (PT) ≤1.5×ULN;
9. Activated partial thromboplastin time (APTT) ≤1.5×ULN. 11.Patients with reproductive capacity, both male and female, must use reliable contraceptive measures during the study medication use and for 60 days after the last dose.

Exclusion Criteria:

* Here is the translation of the provided text into English:

  1. Pathologically diagnosed as a mixed type of hepatocellular carcinoma-intrahepatic cholangiocarcinoma (HCC-ICC).
  2. Positive surgical margins or tumor rupture.
  3. Reoperation for recurrent liver cancer.
  4. History of other malignancies within 5 years, unless the patient has undergone potentially curative treatment and has no evidence of the disease for 5 years, except for patients who have successfully undergone resection surgery for skin basal cell carcinoma, skin squamous cell carcinoma, superficial bladder cancer, cervical carcinoma in situ, or other carcinoma in situ (the 5-year requirement does not apply).
  5. Past or current congenital or acquired immunodeficiency diseases.
  6. Patients who have undergone allogeneic transplantation.
  7. Insufficient biopsy and/or surgical samples are unavailable.
  8. Pregnant and breastfeeding patients.
  9. Received targeted drug therapy such as sorafenib, lenvatinib, regorafenib, or immunomodulatory therapy such as anti-PD-1, anti-PD-L1, anti-CTLA-4 before surgery.
  10. Unable to provide informed consent (due to language, intellectual capacity, etc.).
  11. Active bleeding or coagulation abnormalities, with a tendency to bleed or currently undergoing thrombolytic, anticoagulant, or antiplatelet therapy.
  12. History of gastrointestinal bleeding within the past 4 weeks or a clear tendency towards gastrointestinal bleeding (e.g., known active local ulcer lesions, fecal occult blood ++ or more, if persistent fecal occult blood +, gastroscopy should be performed), or other conditions that may cause gastrointestinal bleeding as determined by the investigator (e.g., severe gastric fundus/esophageal varices).
  13. Significant clinically meaningful cardiovascular diseases, including but not limited to acute myocardial infarction, severe/unstable angina, or coronary artery bypass grafting within the past 6 months, congestive heart failure (New York Heart Association NYHA class >2), arrhythmias that are poorly controlled or require pacemaker treatment, uncontrolled hypertension with medication (systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg).
  14. Allergy to chemotherapy drugs or contraindications to surgery.
  15. History of thrombosis or thromboembolic events within the past 6 months, such as stroke and/or transient ischemic attack, deep vein thrombosis, pulmonary embolism, etc.
  16. History of gastrointestinal perforation, abdominal fistula, or intra-abdominal abscess within the past 6 months.
  17. Not yet recovered from surgery, such as having unhealed incisions or severe postoperative complications.
  18. History of alcohol, psychotropic drugs, or other drug abuse within the past 6 months.
  19. Presence of other serious diseases that the investigator deems unsuitable for participation in this study;
  20. Currently participating in other therapeutic/interventional clinical trials.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
1-year cumulative recurrence-free patient percentage | The patient started taking lenvatinib after radical surgery for hepatocellular carcinoma and continued treatment for up to 1 year.
  Proportion of patients with high-risk recurrent hepatocellular carcinoma who are free of tumor recurrence within one year after curative surgery.

SECONDARY OUTCOMES:
Recurrence Free Survival | The patient started taking lenvatinib after radical surgery for hepatocellular carcinoma and continued treatment for up to 3 years.
  The time elapsed from the date of enrollment to tumor recurrence or death from any cause (if the subject died before disease recurrence). Surviving subjects without confirmed tumor recurrence at the database cutoff date were censored based on the date of the last imaging tumor assessment. The date of tumor recurrence was the date of the first imaging confirmation of tumor recurrence.
Overall Survival | The time span from the date of surgery to the date of the patient's last follow-up visit or death, assessed up to 3 years.
  The elapsed time from the date of enrollment to the date of death from any cause. If the subject was still alive at the database cutoff date, the subject was censored at the date of the last survival follow-up in the database.
Time To Recurrence | The time span from the date of radical liver resection to the date of first documented tumor recurrence, assessed up to 3 years.
  The time elapsed from the date of enrollment to the date of tumor recurrence. Subjects who did not experience tumor recurrence at the database cutoff date were censored at the date of last imaging tumor assessment.
Diachronic changes in quality of life scores based on FACT-Hep scale | From enrollment date to database deadline, assessed up to 3 years.
  The FACT-Hep scale is a 46-item, self-assessed, multidimensional, validated questionnaire used to assess health-related quality of life in subjects with liver cancer types. FACT-Hep assessment dimensions include physical status, social/family status, emotional status, functional status and additional symptoms of hepatocellular carcinoma. Subjects responded to each item on the scale on a scale from 0 (not at all) to 4 (extremely). The average time required to complete the questionnaire is less than 10 minutes. Five subscale scores and one overall score can be calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
Involving patient privacy and biometric information security